CLINICAL TRIAL: NCT00941434
Title: Community Based Management of Malnutrition. A Proposal for Pakistan Initiative for Mothers and Newborns
Brief Title: Community Based Management of Malnutrition
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aga Khan University (Other)
Collaborators: John Snow, Inc. (Industry); Pakistan Ministry of Health (Other Government)
Responsible Party: Prof. Zulfiqar A Bhutta, Aga Khan University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1227-Ped/ERC-09
Record Dates: First submitted 2009-07-16; First posted 2009-07-17 (Estimated); Last update posted 2011-07-08 (Estimated); Status verified 2009-07

CONDITIONS: Severe and Moderate Malnutrition
Keywords: RUTF; SAM; Nutributter

ARMS (1):
- RUTF (Experimental): Children with Severe malnutrition will be treated with Ready to use therapeutic food (RUTF) till their weight for age z scores are no longer in severe malnutrition group
  Interventions: Dietary Supplement: RUTF

INTERVENTIONS:
Dietary Supplement: RUTF — Children with severe malnutrition will be treated with a daily dose of RUTF till their weight for age z scores no longer fall in severe malnutrition group

SUMMARY:
Malnutrition is the leading cause of death in children in developing countries, especially Pakistan. According to World Health Organization about 60% of all deaths, occurring among children aged less than five years in developing countries, could be attributed to malnutrition.

Community-based therapeutic care attempts to maximize population-level impact through improved coverage, access, and cost-effectiveness of treatment. Such community-based nutrition packages can provide effective care to the majority of acutely malnourished children as outpatients, using techniques of community mobilization to engage the affected population and maximize coverage and compliance. Children with SAM without medical complications are treated in an outpatient therapeutic program with ready-to-use therapeutic food and routine medications.

The Ready-to-use Therapeutic Food (RUTF) and Fortified Supplementary food has revolutionized the treatment of moderate and severe malnutrition. The advantage of these commodities is that they are ready-to-use paste which does not need to be mixed with water, thereby avoiding the risk of bacterial proliferation in case of accidental contamination.

DETAILED DESCRIPTION:
Aim:

To evaluate the effectiveness of Ready to Use Therapeutic food and food supplement (Nutributter) in the treatment of Moderate and Severe malnutrition in rural Pakistan when administered at community level

Primary objectives:

* To assess the acceptability, feasibility and effectiveness of Nutributter and Fortified supplementary food (RUTF) in the treatment of moderate malnutrition in children less than three years of age in community settings.
* To assess the acceptability, feasibility and effectiveness of RUTF in the treatment of severe malnutrition in children less than three years of age in community settings.

Methodology:

Study Design: Community based, step wedge randomized trial

Sample size estimation:

Total Population of the study area: 60268. Estimated under 5 years of age Population: 9040 (Assuming 15% of Total population. Estimated Population between 6 months to 3 years: 4520 (Assuming 50% of Under 5 Population)

Sample Size for Moderate Malnutrition:

It is estimated that the Prevalence of Moderately Malnourished: 20% Therefore 20% of 4520: 904. We anticipate recruiting 1000 cases (96 about 10% extra for any loss to follow-ups or drop outs)

Sample Size For Severe Malnutrition:

It is estimated that the prevalence of Severe Acute Malnutrition is 8%. Therefore 8% of 4520: 360. We anticipate recruiting 400 cases (40 about 10% extra for any loss to follow-ups or drop outs)

ELIGIBILITY:
Inclusion Criteria:

* Born and eligible for inclusion within the study period.
* Presence of moderate to severe malnutrition.
* Ability of the parents or guardians to provide informed consent

Exclusion Criteria:

* Presence of chronic debilitating illness.
* Residence outside of study areas.
* Inability or refusal of the parents or guardians to give informed consent, or refusal of assessment.

Ages: 6 Months to 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 800 (Actual)
Dates: Start 2009-07; Primary Completion 2010-06 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Improved Growth Parameters Weight for Age Z Scores. | 1 year

SECONDARY OUTCOMES:
Reduction in Malnutrition related morbidity and mortality patterns in early childhood | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Zulfiqar A. Bhutta, MBBS, FRCP, FCPS, PhD, Principal Investigator — Women and Child Health Division, Aga Khan University
Locations (1):
- AKU Project Office, Dadu, Sindh, Pakistan